CLINICAL TRIAL: NCT06885970
Title: The Effect of Cytisine Treatment for Smoking Cessation on Cardiovascular Function in Adult Smokers of Conventional Combustible Cigarettes and New Tobacco Products-Observational Study.
Brief Title: The Effect of Cytisine Treatment for Smoking Cessation on Cardiovascular Function in Adult Smokers
Acronym: Cytisin-angio
Status: Recruiting | Type: Observational
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Ignatios Ikonomidis, Professor of Cardiology, University of Athens
Other Study IDs: Cytisine_Attikon
Record Dates: First submitted 2025-03-13; First posted 2025-03-20 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Smoking Cessation; Arterial Stiffness; Endothelial Dysfunction
Keywords: arterial stiffness; smoking cessation; myocardial deformation; endothelial glycocalyx
MeSH Terms: conditions — Smoking Cessation | interventions — Nicotine Replacement Therapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Standard dose Cytisine Regime: At least 50 participants will receive cytisine at the standard dose regime [From the 1st to the 3rd day, 1 tablet every 2 hours, 6 tablets; From the 4th to the 12th day, 1 tablet every 2.5 hours, 5 tablets; From the 13th to the 16th day, 1 tablet every 3 hours, 4 tablets; From the 17th to the 20th day, 1 tablet every 5 hours, 3 tablets; From the 21st to the 25th day, 1-2 tablets per day, up to 2 tablets
  Interventions: Drug: Cytisinicline administration
- Nicotine Replacement Therapy: At least 50 participants will receive 50 nicotine replacement therapy
  Interventions: Drug: Cytisinicline administration
- Prolonged Cytisine Regime: A least 50 participants will receive the prolonged cytisine regime (3mg cytosine 3 times daily for 12 weeks
  Interventions: Drug: Cytisinicline administration
- Control Group: At least 50 participants who will not be eager to cease smoking
  Interventions: Drug: Cytisinicline administration

INTERVENTIONS:
Drug: Cytisinicline administration — Participants will receive in the smoki
  Other Names: Nicotine Replacement Therapy

SUMMARY:
Introduction: Pharmacological interventions can enhance smoking cessation success and long-term abstinence. Cytisine, a plant derived alkaloid, is a selective partial agonist at alpha-4 beta-2 nicotinic acetylcholine receptors, which are crucial in nicotine dependence.

Aim of the Study The primary objective of this observational study is to evaluate the efficacy of cytisine in a standard 25-day dosing regimen among adult smokers and users of alternative nicotine products (e-cigarettes or heated tobacco). The study will assess the impact of cytisine on cardiovascular function, including arterial stiffness, cardiac deformation, and endothelial glycocalyx integrity.

The secondary aim is to determine relapse rates post-treatment, treatment side effects, and new cardiovascular events during the treatment period and at six-month follow-up.

Materials and Methods: This observational study will recruit smokers visiting the smoking cessation unit at the 2nd Department of Cardiology, Attikon University Hospital, Athens. All participants will receive counseling and treatment from the attending physician.

A minimum of 200 participants will be enrolled, categorized into:

• At least 50 receiving cytisine in the standard dosing regimen: Days 1-3: 1 tablet every 2 hours (6 tablets daily) Days 4-12: 1 tablet every 2.5 hours (5 tablets daily) Days 13-16: 1 tablet every 3 hours (4 tablets daily) Days 17-20: 1 tablet every 5 hours (3 tablets daily) Days 21-25: 1-2 tablets daily

* At least 50 receiving nicotine replacement therapy
* At least 50 receiving prolonged cytisine therapy (3 mg, three times daily for 12 weeks)
* At least 50 who do not intend to quit smoking (control group)

Assessments will be conducted at baseline, one month, and six months post-recruitment. The following measurements will be performed:

A. Arterial Stiffness: Pulse wave velocity (cf-PWV) using the Complior device to measure arterial stiffness, Augmentation index and pulse wave velocity using the Arteriograph device via brachial artery cuff.

B. Endothelial Glycocalyx Integrity: Perfused boundary region (PBR) assessment of sublingual microvasculature using a Sidestream Dark Field (SDF) camera.

C. Cardiac Function: Left ventricular ejection fraction (LVEF), myocardial strain (GLS), and myocardial work assessment via speckle-tracking echocardiography (Echopac 203, GE Horten Norway).The investigators will also calculate myocardial work (MW) using pressure-strain loop analysis.

D. Oxidative Stress: Plasma malondialdehyde (MDA) and protein carbonyl (PC) levels measured via spectrophotometry.

E. Smoking Cessation Monitoring: Exhaled carbon monoxide (CO) measured using a commercial device (Smokelyzer, Bedfont Scientific Ltd.).

This study aims to provide valuable insights into cytisine's effectiveness in smoking cessation and its impact on cardiovascular health.

DETAILED DESCRIPTION:
Introduction Undoubtedly, smoking is one of the most important risk factors for cardiovascular diseases and smoking cessation is one of the most effective interventions for both primary and secondary prevention. Pharmacological interventions provided accurately can increase the likelihood of both smoking cessation and abstinence long term. Cytisine is a plant alkaloid product that can be isolated from parts of many plant species, mainly from Laburnum seeds.

Cytisine acts as a selective partial agonist at alpha-4 beta-2(acetylcholine) nicotinic receptors which play an important role in nicotine dependence. Its mode of action is very similar to varenicline, a drug already used as an effective way to quit smoking.

Aim of the study The primary objective of this observational study is to study the efficacy of cytisine treatment in the standard dosing regimen in 25 days of treatment in adult smokers and users of alternative nicotine intake products (e-cigarettes or heated cigarettes) with respect the effect of cytisine treatment on cardiovascular function. Cardiovascular function will be addressed by markers of arterial stiffness, cardiac deformation and integrity of the endothelial glycocalyx.

The secondary aim of the study is to assess the degree of relapse to smoking after treatment, the side effects of the treatment and new cardiovascular events during the treatment period and at 6 months follow-up.

Material and Method The present observational study will include smokers who have visited the smoking cessation unit of the 2nd Department of Cardiology, Attikon University Hospital, Athens. All participants are receiving guidance and treatment by the attending physician of the smoking cessation Unit.

The investigators are planning to include at least 200 individuals, out of which: at least 50 will receive cytisine at the standard dose regime [From the 1st to the 3rd day, 1 tablet every 2 hours, 6 tablets; From the 4th to the 12th day, 1 tablet every 2.5 hours, 5 tablets; From the 13th to the 16th day, 1 tablet every 3 hours, 4 tablets; From the 17th to the 20th day, 1 tablet every 5 hours, 3 tablets; From the 21st to the 25th day, 1-2 tablets per day, up to 2 tablets], at least 50 are on nicotine replacement therapy , at least 50 who will receive the prolonged cytisine regime (3mg cytisine 3 times daily for 12 weeks) and at least 50 that are not eager to quit smoking, as a control group.

Exclusion criteria are: history of coronary artery disease, active malignancy, history of severe liver and renal failure, history of autoimmune disease. After being informed in detail and signing the required consent forms, smokers will be asked to complete specific questionnaires on nicotine dependence (Fagerstrom Test) and depression (Zung score). A complete history on their smoking habits, medical history, demographic and socio-economic characteristics will also be obtained.

Assessment will be performed at baseline, at 1 month and at 6 months post recruitment.

All participants of the study will the following measurements in each assessment:

A. Measurement of pulse wave velocity, (cf-PWV) with the complior device (Complior, Alam Medical, Vincennes, France) by applying two sensors to the common carotid and femoral artery as a metric of arterial stiffness. Carotid-to-femoral PWV is the ratio of the distance between the carotid and femoral pulse palpation site to the pulse wave transit time (m/s).

Β. Calculation of the pulse wave velocity and the pulse wave amplification index (aorta augmentation index) with the arteriograph device, by applying a cuff to the brachial artery .

C. The investigators will evaluate the perfused boundary region (PBR, μm) of the sublingual microvasculature utilizing Sidestream Dark Field (SDF) camera (Microscan, GlycoCheck, Microvascular Health Solutions Inc., Salt Lake City, UT, USA) with diameter range 4 to 25 μm. SDF camera implements green reflected light emitting diode (LED) light (540 nm) to depict the hemoglobin in red blood cells (RBCs) . The camera is placed under the tongue and captures over 3000 microvessels segments. The valid captured images (those with good focus, good contrast, and minimal level of tissue motion) are saved and analyzed by the GlycoCheck software . The median RBC column width and the total perfused diameter of the microvessels are assessed by the software. PBR is estimated by the formula: (perfused diameter-median RBC column width)/2 . Afterwards the software calculates the PBR of the microvessels with diameter ranging from 4-9 μm, 10-19 μm and 20-25 μm . High PBR imply that RBCs penetrate more deeply into the endothelial surface which represents a compromised glycocalyx layer with affected barrier properties and vice versa. The measurement takes approximately three minutes to complete. The reported variability for PBR calculation of the same and between different observers are 4.3% and 5.2%, respectively. Of note, PBR evaluation is independent of hematocrit, as the software encompasses solely vessel segments with red blood cells filling percentage of more than 50% .

D. In addition, cardiac function will be assessed by calculating left ventricular ejection fraction (LV), myocardial strain (GLS) and myocardial work (myocardial work) using the spreckle tracking echocardiography. Myocardial deformation was assessed by way of 2-dimensional strain measurement, with speckle-tracking analysis by dedicated software (Echopac 203, GE Horten Norway). LV apical 2-, 3-, and 4-chamber views at ≥50 frames per second frame rate were acquired and the global longitudinal strain (GLS) is calculated from the respective apical views, applying previously published methodology. PWV/ GLS ratio (-m/s %) was calculated as a marker of ventricular arterial interaction. Myocardial work (MW) wil be estimated by combining echo-derived left ventricular (LV) strain with brachial blood pressure to construct LV strain-pressure curves non-invasively. Brachial cuff systolic pressure measurements provide the peak systolic LV pressure value, which is combined with the input of valvular timing events that define isovolumetric and ejection phases, allowing the construction of an LV pressure curve. This is combined with LV strain data into a pressure-strain loop (PSL), the area within which represents MW. Global MW index (GWI) is defined as the work within the LV PSL from mitral valve closure to mitral valve opening, while constructive MW (GCW) is the component of MW that contributes to LV ejection. On the contrary, wasted MW (GWW) is the work wasted as myocyte lengthening during systole, which does not contribute to LV ejection. MW efficiency (GWE) is defined as the ratio of GCW to the sum of GCW and GWW [GWE=GCW/(GCW+GWW)].

E. Oxidative stress. A commercially available spectrophotometry kit (Oxford Biomedical Research, Rochester Hills, Mich, colorimetric assay for lipid peroxidation; measurement range 1-20 nmol/l) was used to determine plasma MDA levels. Plasma PC levels will be measured by spectrophotometrical assessment of 2,4-dinitrophenylhydrazine PC derivatives and results are expressed as nmol/mg protein. For MDA and PC, the intra-assay variability is 3.39% and 4.52%, respectively and the inter-assay variability is 4.75% and 5.93%, respectively.

F. Exhaled CO will also be measured using a commercial device (Smokelyzer, Bedfont® Scientific Ltd Station Road).

Statistical analysis Statistical analysis will be conducted by SPSS version 29 (IBM SPSS Statistics, Inc., Chicago, IL, USA). All scale variables are presented as mean ± SD in case of normal distribution. The normality tests Kolmogorov-Smirnov and Shapiro-Wilk will be applied to determine the distribution. When normality criteria are not met, the investigators will transform the variables into ranks. Categorical variables will be presented as absolute and relative frequencies. The investigators will perform Spearman or Pearson correlation tests, as appropriate, for correlation analysis. Nominal variables are examined using either Chi-square tests or Fisher's exact tests, as appropriate. Analysis of Variance (ANOVA) for repeated measurements will be implemented for comparisons between and within subjects regarding cardiovascular parameters and smoking status. The F and the corresponding p values for the change of the markers at follow up measurement are estimated. Also, the F and p values for the effect between time of measurement and the intervention arms will be calculated. When Mauchly's test indicated that the sphericity assumption is not satisfied, corrections such as Greenhouse-Geisser, Huynh-Feldt, or Lower-Bound are applied. All statistical tests are two-tailed, with a p-value of less than 0.05 deemed statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Smokers willing to participate

Exclusion Criteria:

* history of coronary artery disease, active malignancy, history of severe liver and renal failure, history of autoimmune disease.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: We are planning to include at least 200 smokers individuals, out of which: at least 50 will receive cytisine at the standard dose regime [From the 1st to the 3rd day, 1 tablet every 2 hours, 6 tablets; From the 4th to the 12th day, 1 tablet every 2.5 hours, 5 tablets; From the 13th to the 16th day, 1 tablet every 3 hours, 4 tablets; From the 17th to the 20th day, 1 tablet every 5 hours, 3 tablets; From the 21st to the 25th day, 1-2 tablets per day, up to 2 tablets], at least 50 are on nicotine replacement therapy , at least 50 who will receive the prolonged cytisine regime (3mg cytosine 3 times daily for 12 weeks) and at least 50 that are not eager to quit smoking, as a control group.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2025-07-22 (Estimated); Study Completion 2025-08-10 (Estimated)

PRIMARY OUTCOMES:
Comparisons of changes in arterial stiffness between treatment groups | 0, 1, 6 months
  Comparisons of changes in carotid-to-femoral Pulse Wave Velocity between treatment groups
Comparisons of changes in endothelial glycocalyx integrity between treatment groups | 0,1, 6 months
  Comparisons of changes in Perfused Boundary Region of sublingual microvessels with diameter range 4-25 μm.
Comparisons of changes in myocardial performance between treatment groups | 0,1, 6 months
  Changes in Global Longitudinal Strain of the Left Ventricle via echocardiography beween treatment groups

SECONDARY OUTCOMES:
Comparisons of changes in oxidative stress burden between treatment groups | 0,1,6 months
  Comparisons of changes in Malondialdehyde levels between treatment groups
Comparisons of changes in smoking cessation rates between treatment groups | 0,1,6 months
  Comparisons of changes exhaled Carbon Monoxide levels between treatment groups

CONTACTS AND LOCATIONS:
Locations (1):
- Attikkon University Hospital, Athens, Haidari, Greece